CLINICAL TRIAL: NCT02110121
Title: Picosure Alexandrite Laser and Revlite Nd:Yag Laser for the Treatment of Unwanted Tattoos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PICOREVLITE
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Unwanted Tattoos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Picosure Laser System (Experimental): Picosure Laser System for the Treatment of Unwanted Tattoos
  Interventions: Device: Picosure Laser System
- Revlite Laser System (Experimental): Revlite Laser System for the Treatment of Unwanted Tattoos
  Interventions: Device: Revlite Laser System

INTERVENTIONS:
Device: Picosure Laser System — Picosure Laser System for the Treatment of Unwanted Tattoos
  Arms: Picosure Laser System
Device: Revlite Laser System — Revlite Laser System for the Treatment of Unwanted Tattoos
  Arms: Revlite Laser System

SUMMARY:
The purpose of this study is to evaluate the Picosure and Revlite Laser Systems for the treatment of unwanted tattoos.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy non-smoking (must have quit 6 months prior) male or female between 18 and 65 years old.
2. Is willing to consent to participate in the study.
3. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitizing medication.
3. The subject has active or localized systemic infections.
4. The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy {greater than 81 mg per day}).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. The subject has used Accutane within 6 months prior to enrollment.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has a history of keloid scar formation.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of basal cell carcinoma, squamous cell carcinoma or melanoma.
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications or has an autoimmune disorder.14. The subject has red tattoo ink allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Cynosure Inc., Westford, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Picosure Laser System | Revlite Laser System
Started | 58 | 5
Completed | 42 | 5
Not Completed | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Picosure Laser System | Revlite Laser System | Total
Number analyzed (Participants) | 58 | 5 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 5 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 3 | 34
  Male | 27 | 2 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 51 | 5 | 56
  Race/Ethnicity: Hispanic | 5 | 0 | 5
  Race/Ethnicity: Asian | 2 | 0 | 2
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 2 | 0 | 2
    Fitzpatrick Skin Type II | 17 | 1 | 18
    Fitzpatrick Skin Type III | 31 | 4 | 35
    Fitzpatrick Skin Type IV | 5 | 0 | 5
    Fitzpatrick Skin Type V | 2 | 0 | 2
    Fitzpatrick Skin Type VI | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Clearance
Description: Clearance will be measured using a blinded photograph evaluation scale. This ranges from 0 to 3, where a score of 0 is 0-25%, 1 is 25-50% clearance rating, 2 is 50-75%, and 3 is >75%. Photographs will be taken of the subjects at baseline and post treatment. The results will be compared to determine clearance.
Time Frame: 2 months post each patient's last treatment, approximately 15 months
Population: 11 Picosure subjects were lost to follow up, 2 subjects withdrew, and 7 subjects were not required to attend the follow up because the study was ended.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: tattoos
Arm/Group | Picosure Laser System | Revlite Laser System
Number analyzed (Participants) | 43 | 5
Number analyzed (tattoos) | 81 | 5
score on a scale | 2.5 (.7) | 3.0 (0.0)

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected for each patient's participation in the study, about 15 months. Adverse events that are not resolved by this time will be followed up with until the condition resolves, stabilizes, or is otherwise explained, or the subject is lost to follow-up.
Arm/Group | Picosure Laser System | Revlite Laser System
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/5
Other Adverse Events (participants affected / at risk) | 45/58 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Picosure Laser System (N=58) | Revlite Laser System (N=5)
Edema (Skin and subcutaneous tissue disorders) | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0
Pinpoint Bleeding (Skin and subcutaneous tissue disorders) | 26 | 5
Bruising (Skin and subcutaneous tissue disorders) | 2 | 0
Blistering (Skin and subcutaneous tissue disorders) | 10 | 1
Redness (Skin and subcutaneous tissue disorders) | 23 | 4
Swelling (Skin and subcutaneous tissue disorders) | 17 | 3
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Other (Skin and subcutaneous tissue disorders) | 2 | 2
Scabs (Skin and subcutaneous tissue disorders) | 3 | 0
Purpura (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT02110121/SAP_000.pdf
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02110121/Prot_001.pdf